CLINICAL TRIAL: NCT03896906
Title: Comparison of Preoxygenation With a High-flow Nasal Cannula and a Simple Mask Before Intubation During Induction of General Anesthesia in Patients Undergoing Head and Neck Surgery
Brief Title: Preoxygenation With a High-flow Nasal Cannula or a Simple Mask Before General Anesthesia in Head and Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Soo Choi, MD, PhD, Assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0275
Record Dates: First submitted 2019-03-06; First posted 2019-04-01 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Neoplasm
Keywords: preoxygenation; high-flow nasal cannula
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group N (Experimental): pre-oxygenation with High-flow nasal cannula
  Interventions: Device: High-flow nasal cannula
- Group M (Active Comparator): pre-oxygenation with simple mask
  Interventions: Device: simple mask

INTERVENTIONS:
Device: High-flow nasal cannula — Apply high ﬂow heated (34 °C) and humidified nasal oxygen with the OptiFlow System (Thrive, Fisher & Paykel®, Aukland New Zealand) using a ﬂow of 30 liter/minute and an inspiratory oxygen fraction (FiO2) of 1.0. Increase the oxygen flow to 60 liter/minute over the course of the first minute. Ask the patients not to speak during anesthesia induction and keep the mouth closed.
  Arms: Group N
Device: simple mask — Perform standard preoxygenation by oxygen insufflation via a face mask using the standard anesthesia ventilators (semicircular system) with 100% oxygen ﬂow of 12 liter/minute. The patients breathe with tidal volume.
  Arms: Group M

SUMMARY:
Objectives: To assess arterial oxygen partial pressure (PaO2) at defined time points during the preoxygenation and to compare between high ﬂow heated humidified nasal oxygen versus standard preoxygenation with oxygen insufflation via face mask over at least 5 minutes Methods: This randomized, single-blinded, prospective study was conducted at Asan Medical Center in Seoul, Republic of Korea.

Populations: Patients undergoing head and neck surgery Expected outcomes: The course of PaO2 levels is superior to those of the face mask during the whole preoxygenation procedure and after the intubation.

DETAILED DESCRIPTION:
Rationale & background information:

Pre-oxygenation before general anesthesia is usually achieved using oxygen delivered via a facemask before induction of anesthesia; this potentially extends the time available for securing the airway before hypoxemia to 6 min. The lungs are commonly ventilated with a bag/facemask technique after induction, and this can be repeated if attempts at intubating the trachea are prolonged. However, facemask ventilation has traditionally been avoided in the circumstance which has the risk of gastric insufflation of gas, leading to increased intragastric pressure and raised risk of pulmonary aspiration of stomach contents. In addition, if difficult ventilation is anticipated, facemask ventilation may not be possible at all, and 6 minutes with hypoxemia may be insufficient for intubation.

An ideal preoxygenation to extend apnea tolerance during anesthesia induction is essential to avoid live threatening airway incidents. The high-flow nasal cannula, the OptiFlow System (Thrive, Fisher & Paykel®, Aukland New Zealand), has the ability to deliver warmed and humidified oxygen through specially designed nasal cannula and enable oxygen to be comfortably delivered at rates of > 70 liter/min. Several study showed that nasal delivery of humidified oxygen to paralyzed and anesthetized patients at these rates maintains oxygenation and achieves acceptable carbon dioxide concentration. The investigators hypothesized that an extended apneic period without facemask ventilation could be particularly beneficial to patients undergoing general anaesthesia.

Study goals and objectives:

To assess arterial oxygen partial pressure (PaO2) at defined time points during the preoxygenation and to compare between high ﬂow heated humidified nasal oxygen versus standard preoxygenation with oxygen insufflation via face mask over at least 5 minutes

ELIGIBILITY:
Inclusion Criteria:

1. Patients with head and neck cancer undergoing resection surgery planned arterial cannulation and invasive arterial blood pressure monitoring and arterial blood gas analysis
2. Patients over 19-year old
3. Patients who voluntarily participated in the study
4. Patents in American Society of Anesthesia physical status 1-3

Exclusion Criteria:

1. Patients who don't approve to participation
2. Unable to give informed consent because of a language barrier
3. Patients with severe respiratory disease
4. Patients with severe cardiovascular or cerebrovascular disease
5. Patients with severe psychiatric disorders
6. Anyone who is not appropriate according to researcher's decision

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
PaO2 (arterial oxygen partial pressure) at pre-defined time points. | through study completion, an average of 10 minutes
  changes of PaO2

SECONDARY OUTCOMES:
degree of blood oxygenation oxygenation | through study completion, an average of 10 minutes
  result of arterial blood gas analysis
various patients' characteristics about airway | through study completion, an average of 10 minutes
  upper lip bite test classification (class 1~3)
degree of difficulty for intubation | through study completion, an average of 10 minutes
  the number of attempts at laryngoscopy and use of any rescue maneuvers, seniority of the anesthesiologist
degree of tissue oxygenation | through study completion, an average of 10 minutes
  O2 saturation

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Soo Choi, Dr., Principal Investigator — Department of Anesthesiology and Pain Medicine, Asan Medical Center
Locations (1):
- Jun-Young Jo, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jo JY, Kim WJ, Ku S, Choi SS. Comparison of preoxygenation with a high-flow nasal cannula and a simple mask before intubation during induction of general anesthesia in patients undergoing head and neck surgery: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Mar;99(12):e19525. doi: 10.1097/MD.0000000000019525. PMID 32195955